CLINICAL TRIAL: NCT06233812
Title: Surgical Outcomes of Simple Interrupted Versus Running Epidermal Sutures in Full-thickness Skin Graft Placement: A Split-scar, Randomized, Non-inferiority Comparison
Brief Title: Surgical Outcomes of Simple Interrupted Versus Running Epidermal Sutures in Full-thickness Skin Graft Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 23-0413
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Skin Graft Scar

STUDY DESIGN:
Intervention Model Description: Patients will serve as their own controls -- one half of the full-thickness skin graft will be sutured with simple running sutures and the other half with simple interrupted sutures.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half A of the FTSG (Active Comparator): "A" (superior or left relative to the patient, depending on the shape of the wound)
  Interventions: Procedure: Simple interrupted suturing technique; Procedure: Running suturing technique
- Half B of the FTSG (Active Comparator): "B" (inferior or right relative to the patient).
  Interventions: Procedure: Simple interrupted suturing technique; Procedure: Running suturing technique

INTERVENTIONS:
Procedure: Simple interrupted suturing technique — Both simple interrupted and running epidermal sutures are considered acceptable, appropriate techniques for FTSG placement. Therefore, this study would be important in determining whether running sutures, the more efficient method, are non-inferior to simple interrupted sutures.
Procedure: Running suturing technique — Both simple interrupted and running epidermal sutures are considered acceptable, appropriate techniques for FTSG placement. Therefore, this study would be important in determining whether running sutures, the more efficient method, are non-inferior to simple interrupted sutures.

SUMMARY:
The study hypothesis is that the use of running epidermal sutures in full-thickness skin graft (FTSG) placement for patients undergoing dermatologic surgery (Mohs micrographic surgery or excision) is non-inferior to the use of simple interrupted sutures with respect to cosmetic outcome. This will be a split-scar (within-person) study, in which half of each participant's scar will receive the study intervention (running epidermal sutures), with the other half receiving the control intervention (simple interrupted sutures). The primary outcome, total observer score of the Patient and Observer Scar Assessment Scale (POSAS) 2.0, will be assessed by two blinded observers at a 3-month follow-up visit, and compared between scar halves.

DETAILED DESCRIPTION:
A FTSG is used in lieu of linear repair or local tissue skin flap rearrangement when surrounding skin tissue laxity is unavailable or the patient prefers a graft instead. Typically the skin for a FTSG is harvested from a local or distant donor site depending on skin tissue match and tissue availability and sutured into place. The site where the FTSG was taken is primarily repaired or allowed to heal via second intent. This study is important because it provides a comparison of cosmetic outcome between interrupted versus running cutaneous sutures. The information provided would help determine if a more efficient suturing technique is non-inferior to a less efficient one, thus saving time for the patient and provider. There is no current standard of practice, with dermatologic surgeons using both interrupted and running sutures, as there is a paucity of literature on this topic as related to full thickness grafts after dermatologic surgery. Running epidermal sutures are more time efficient and thus decrease patient intra-operative time, save on suture material, increase surgeon productivity, and may improve the overall patient operative experience. There have been multiple other split scar studies and studies related to the cosmetic outcomes of various suturing practices. However, there have been none that have looked at simple versus running epidermal stitching of FTSG placement.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will capture patients
* 18 years or older
* have a FTSG reconstruction
* any body site
* to close to a primary defect after dermatologic surgery.

The authors will exclude patients not undergoing reconstruction with full-thickness skin-graft placement, unable to return for follow-up visits, unable to provide consent (eg. unable to understand spoken/written English, mentally handicapped), and patients under 18 years of age. Male and female patients are eligible. Planned enrollment based on a priori sample size calculation is 52 patients.

Exclusion Criteria:

* Not undergoing reconstruction with full-thickness skin-graft placement
* FTSG not large enough to accommodate at least 3 interrupted sutures on one half side
* Pregnancy or lactation
* Under 18 years of age
* Unable/unwilling to return for follow-up visits
* Unable to provide consent (eg. unable to understand spoken/written English, mentally handicapped)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The Patient and Observer Scar Assessment Scale (POSAS) | POSAS 2.0 observer total score at 3 months post-surgery, calculated as the average of two observers' total scores.
  Total observer score of the Patient and Observer Scar Assessment Scale (POSAS) 2.0
  The patient score combines scar pain, itch, color, stiffness, thickness, and irregularity (1-10). The observer scale comprises of the items vascularity, pigmentation, thickness, relief, pliability, and surface area. All items of the patient and observer score combined will form a total POSAS score (the highest score represents the worst scar imaginable). It also consists of an overall opinion of the scar

SECONDARY OUTCOMES:
Clinician overall opinion | through study completion, an average of 1 year
  Clinician observer overall opinion of scar quality, measured on a 10-point scale (1-10) by two observers and averaged
Patient overall opinion | through study completion, an average of 1 year
  Patient overall opinion of scar quality, measured on a 10-point scale (1-10)
Complications | through study completion, an average of 1 year
  Number of patients experiencing bleeding requiring physician intervention after surgery Number of patients experiencing graft failure Number of patients developing infection between date of surgery and 3-month follow-up visit Number of patients with hypertrophic or keloidal scar formation Number of patients experiencing wound dehiscence (re-opening) between surgery and the 3-month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Victoria R Sharon, MD, Principal Investigator — Northwell Dermatology
Locations (1):
- Marcus Elias, North New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No